CLINICAL TRIAL: NCT03924180
Title: Glytactin EfficiEncy in Non or Insufficiently Treated Adult PHENylketonuria Patients
Acronym: GLEEPHEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR180127 - GLEEPHEN; 2018-A03244-51 (Registry Identifier: IRCB)
Record Dates: First submitted 2019-04-22; First posted 2019-04-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Adult Phenylketonuria Non Treated Patients
Keywords: Amino acid; GMP; PKU
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled trial performed in open and 2 parallel groups: "GMP" versus "amino acids" group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMP - Dietary Supplement for PKU patients (Experimental): Glycomacropeptides -GMP Glytactin
  Interventions: Dietary Supplement: Dietary Supplement for PKU patients
- Control -Amino acids mixtures (Active Comparator): Mixtures of conventional amino acids.
  Interventions: Dietary Supplement: Dietary Supplement for PKU patients

INTERVENTIONS:
Dietary Supplement: Dietary Supplement for PKU patients — For both treatment groups, the objective in total protein will be 1g / kg / day of ideal weight, in 3-6 doses / day, including natural proteins and supplemented by the products under study.

SUMMARY:
Phenylketonuria is the most common inherited metabolic disease in France and is screened for neonatal exposure. Management consists of a strict and restrictive hypoproteic diet and the intake of amino acid substitutes and dietary supplements free of phenylalanine.One of the major difficulties, which is the source of many treatment failures, is the inappetence of the amino acid supplements required during a strict hypoproteic diet. New formulations, Glycomacropeptides (GMP), have recently appeared and are considered more palatable than conventional amino acid mixtures.

DETAILED DESCRIPTION:
Phenylketonuria is the most common inherited metabolic disease in France and is screened for neonatal exposure. Management consists of a strict and restrictive hypoproteic diet and the intake of amino acid substitutes and dietary supplements free of phenylalanine. If the benefits of treatment are indisputable in children in terms of cognitive prognosis, this benefit is discussed once brain development is complete, especially as many adult patients are no longer treated. However, cognitive, neurological and reversible white matter disorders undergoing treatment are increasingly reported in adult phenylketonurics. As a result, recent European recommendations advocate the maintenance of life-long treatment. One of the major difficulties, which is the source of many treatment failures, is the inappetence of the amino acid supplements required during a strict hypoproteic diet. New formulations, Glycomacropeptides (GMP), have recently appeared and are considered more palatable than conventional mixtures.

PRIMARY OBJECTIVE:

Demonstrate a better metabolic balance under GMP treatment than a conventional amino acid mixture in adult phenylketonuric patients when resuming treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥18 years on an empty stomach
* Phenylketonuric patient Patient with Phenylalaninemia ≥ 900μmol / L on a blotter performed during the screening period (or average of blotter results ≥900 μmol / L if several blotters performed during the screening period)
* Untreated or insufficiently treated patient: not taking or insufficiently Dietary foods for special medical purposes for his PKU, regardless of diet, at the discretion of the investigator
* Patient having signed a free, informed and express consent
* Patient requiring a diet restricted in natural proteins

Exclusion Criteria:

* Protected patient: court bail
* Patient with concomitant diseases / conditions that may compromise the study, at the discretion of the investigator
* Participated in a clinical trial or trial to evaluate PKU foods or treatments in the last 7 days prior to inclusion or planned during the next 6 months
* Participation in an interventional study with health products during the next 6 months
* Pregnancy project within 6 months, pre-conception diet, pregnancy or breastfeeding
* Refusal to consume only validated complements for the protocol
* Phenylketonuria undergoing treatment with BH4
* Allergy to the product under study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Rate of phenylalaninemia on blotter | 6 months
  Rate of phenylalaninemia on blotter measured bi-monthly during the 6 months of the study.

SECONDARY OUTCOMES:
Therapeutic compliance | 6 months
  Therapeutic compliance measured after 3 months and 6 months of treatment
Evolution of neuropsychological tests | 6 months
  Neuropsychological tests measured after 3 months and 6 months of treatment
MRI brain M0, M6 evolution | 6 months
  MRI brain evolution between inclusion and 6 months of treatment
Bone remodeling markers | 6 months
  Bone remodeling markers at inclusion and 6 months of treatment
Evolution of quality of life (PKU QoL score), mood (POMS test - Fillion 1999), at M0, M3, M6. | 6 months
  Evolution of quality of life scores at inclusion, 3 months and 6 months of treatment
Nutritional and clinical markers evaluated at inclusion and 6 months of treatment | 6 months
  Evolution of nutritional and clinical markers at inclusion and 6 months of treatment
Gastrointestinal tolerance at M3 and M6 | 6 months
  Evolution of Gastrointestinal tolerance after 3 months and 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adrien BIGOT, MD-PHD, Study Director — University Hospital of TOURS
Locations (7):
- France (7):
  - CHRU-Hôpital Bretonneau - Service de Médecine Interne-Nutrition, Tours, Centre-Val de Loire
  - CHU-ANGERS -Médecine Interne, Angers
  - CHU du Morvan-Département de Pédiatrie et génétique médicale,, Brest
  - Hôpital Femme-Mère-Enfant-Centre de Référence des Maladies Héréditaires du Métabolisme de Lyon, Bron
  - CHU de LILLE-Hôpital Claude HURIEZ-Service d'Endocrinologie, Lille
  - CHU-Service de Réanimation Pédiatrique / Néonatalogie, Consultation spécialisée en Maladies Héréditaires du Métabolisme, Nantes
  - CHU-RENNES-Hôpital Sud-Service de Génétique-Clinique, Rennes